CLINICAL TRIAL: NCT07332884
Title: Comparison of Mirror Therapy and Routine Physical Therapy for the Management of Pain, Spasticity, and Strength in Patients With Complex Regional Pain Syndrome (CRPS): A Randomized Clinical Trial
Brief Title: Comparative Effects of Mirror Therapy and Standard Physiotherapy in Complex Regional Pain Syndrome
Acronym: (CRPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 70146229@student.uol.edu.pk
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Complex Regional Pain Syndrome
Keywords: Complex Regional Pain Syndrome CRPS; Motor Function; Mirror therapy; Neuro rehabilitation; Pain management
MeSH Terms: conditions — Complex Regional Pain Syndromes; Agnosia | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: This is a parallel-group interventional study in which eligible participants with Complex Regional Pain Syndrome are allocated into two intervention arms. One group receives mirror therapy in addition to routine physical therapy, while the comparison group receives routine physical therapy alone. Participants remain in their assigned intervention group for the duration of the study, and outcomes are assessed at baseline and after completion of the intervention period.
Who Masked: Outcomes Assessor
Masking Description: Masking in a clinical trial refers to the process of concealing certain information from participants, investigators, or other involved parties to prevent bias in the study's outcomes. In addition to the primary parties listed (such as participants, investigators, or outcome assessors), other parties who may be masked can include data analysts, laboratory personnel, or pharmacists responsible for preparing interventions. This ensures that those involved in handling, analyzing, or interpreting study data remain unaware of group assignments, maintaining the integrity and objectivity of the trial results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mirror Therapy Group (Experimental): Participants in this arm will receive mirror therapy, a rehabilitation technique where movements of the unaffected limb are reflected in a mirror to create a visual illusion that the affected limb is moving normally. Therapy sessions will be conducted [specify frequency, e.g., 30 minutes per day, 5 days a week] for [specify duration, e.g., 4 weeks].
  Interventions: Other: Mirror Therapy
- Routine Physical Therapy Group (Experimental): Participants in this arm will receive standard physical therapy for CRPS, including exercises, stretching, and functional activities aimed at improving mobility, reducing pain, and enhancing limb function. Sessions will be conducted [specify frequency, e.g., 30 minutes per day, 5 days a week] for [specify duration, e.g., 4 weeks].
  Interventions: Other: Routine Physical Therapy

INTERVENTIONS:
Other: Mirror Therapy — Participants perform movements with the unaffected limb while watching its reflection in a mirror, creating the visual illusion that the affected limb is moving normally. Aimed at reducing pain and improving motor functio
  Arms: Mirror Therapy Group
Other: Routine Physical Therapy — Standard physical therapy including stretching, strengthening, and functional exercises to improve mobility, reduce pain, and restore limb function in CRPS patients.
  Arms: Routine Physical Therapy Group

SUMMARY:
Complex Regional Pain Syndrome (CRPS) is a chronic pain condition characterized by persistent pain, sensory disturbances, motor dysfunction, and functional impairment, often following trauma or surgery. Conventional physical therapy is commonly used in the management of CRPS; however, treatment outcomes are often variable and incomplete. Mirror therapy is a non-invasive rehabilitation technique that uses visual feedback to influence cortical reorganization and may help reduce pain and improve motor function in patients with CRPS.

The purpose of this study is to compare the effectiveness of mirror therapy with routine physical therapy in patients diagnosed with Complex Regional Pain Syndrome. Eligible participants will be allocated into two groups. One group will receive mirror therapy in addition to standard rehabilitation exercises, while the control group will receive routine physical therapy alone. Both interventions will be delivered over a defined treatment period under supervised conditions.

Primary outcomes will include changes in pain intensity, while secondary outcomes will assess functional ability, range of motion, and overall limb use. Outcomes will be measured at baseline and after completion of the intervention period. This study aims to determine whether mirror therapy provides additional benefits over routine physical therapy in reducing pain and improving functional outcomes in patients with Complex Regional Pain Syndrome.

DETAILED DESCRIPTION:
Complex Regional Pain Syndrome (CRPS) is a disabling chronic pain condition that may develop after injury, surgery, or immobilization and is associated with disproportionate pain, sensory abnormalities, motor dysfunction, and reduced use of the affected limb. These impairments significantly affect daily activities and quality of life. Although routine physical therapy remains a cornerstone of CRPS management, optimal rehabilitation strategies continue to be explored.

Mirror therapy is a neurorehabilitation technique that provides visual feedback of the unaffected limb to create the illusion of normal movement in the affected limb. This approach is believed to modulate central nervous system processing, reduce maladaptive cortical reorganization, and improve motor control. Previous studies have suggested potential benefits of mirror therapy in chronic pain conditions; however, evidence comparing mirror therapy with routine physical therapy in CRPS remains limited.

This study is designed to evaluate and compare the effects of mirror therapy and routine physical therapy on pain and functional outcomes in patients diagnosed with Complex Regional Pain Syndrome. Participants will be assigned to one of two intervention groups. The experimental group will receive mirror therapy sessions alongside conventional rehabilitation exercises, while the control group will receive routine physical therapy based on standard clinical practice. Interventions will be administered by qualified physical therapists according to a predefined treatment protocol.

Outcome assessments will be conducted at baseline and at the end of the intervention period using standardized and validated measures. The study will assess changes in pain intensity, functional performance, and limb use to determine the comparative effectiveness of mirror therapy versus routine physical therapy. Findings from this study may contribute to evidence-based rehabilitation strategies for patients with Complex Regional Pain Syndrome.

ELIGIBILITY:
Inclusion criteria

* Age 40-65 years
* Both genders
* Hemiplegic patients with subacute stage
* Patients who developed CRPS of the hand due to stroke
* Patients with a diagnosis of CRPS 1

Exclusion criteria Cognitive disorders and perceptual disorders

* Comorbid conditions (e.g., decompensated heart failure, chronic renal insufficiency
* Hand arthritis
* Arterial/venous injuries and/ or undergoing arterial revascularization

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Pain management | Duration of intervention: 4 weeks Frequency: 30 minutes per session, 5 sessions per week Pain assessments will be conducted at baseline (pre-intervention), weekly during the intervention, and at the end of 4 weeks to evaluate changes in pain intensity
  Participants in both arms will receive interventions aimed at reducing pain associated with Complex Regional Pain Syndrome. For the Mirror Therapy Group, pain reduction is targeted through visual-motor feedback, which can help retrain the brain and reduce pain perception. For the Routine Physical Therapy Group, pain is managed through exercises, stretching, and functional activities that improve mobility, reduce stiffness, and decrease pain intensity.
Hand Grip | • Baseline assessment: Before the start of the intervention • Interim assessments: Weekly during the 4-week intervention period • Final assessment: At the end of 4 weeks
  Hand grip strength will be measured using a dynamometer to assess the functional strength of the affected limb in patients with Complex Regional Pain Syndrome. Participants will be instructed to squeeze the dynamometer maximally for a few seconds, and the best of three trials will be recorded for accuracy. This measurement evaluates improvements in motor function and muscle strength as a result of the intervention.
spasticity | Baseline: Before the start of the intervention • Interim assessments: Weekly during the 4-week intervention period • Final assessment: At the end of 4 weeks
  Spasticity of the affected limb will be assessed using the Modified Ashworth Scale (MAS), which grades muscle tone from 0 (no increase in tone) to 4 (rigid in flexion or extension). The assessment evaluates resistance to passive movement, helping to determine changes in muscle stiffness and motor control resulting from the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Lahore teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ozdemir EC, Elhan AH, Kucukdeveci AA. Effects of mirror therapy in post-traumatic complex regional pain syndrome type-1: a randomized controlled study. J Rehabil Med. 2024 Sep 24;56:jrm40417. doi: 10.2340/jrm.v56.40417. PMID 39318174
- [Result] Kotiuk V, Burianov O, Kostrub O, Khimion L, Zasadnyuk I. The impact of mirror therapy on body schema perception in patients with complex regional pain syndrome after distal radius fractures. Br J Pain. 2019 Feb;13(1):35-42. doi: 10.1177/2049463718782544. Epub 2018 Jun 13. PMID 30671237
- [Result] Khoramdel F, Ravanbod R, Akbari H. Effect of high-intensity laser therapy and mirror therapy on complex regional pain syndrome type I in the hand area: A randomized controlled trial. J Hand Ther. 2025 Oct-Dec;38(4):791-798. doi: 10.1016/j.jht.2025.02.009. Epub 2025 Mar 21. PMID 40118675
- [Result] Harmsen, W. J., Bulten, R., & Schrier, E. (2020). The effectiveness of mirror therapy and graded motor imagery for complex regional pain syndrome: A randomized controlled trial. European Journal of Pain, 24(8), 1575-1587.
- [Result] Giostri GS, Souza CDA. Complex Regional Pain Syndrome. Rev Bras Ortop (Sao Paulo). 2024 Apr 22;59(4):e497-e503. doi: 10.1055/s-0044-1779331. eCollection 2024 Aug. PMID 39239587
- [Result] Ferraro MC, Cashin AG, Wand BM, Smart KM, Berryman C, Marston L, Moseley GL, McAuley JH, O'Connell NE. Interventions for treating pain and disability in adults with complex regional pain syndrome- an overview of systematic reviews. Cochrane Database Syst Rev. 2023 Jun 12;6(6):CD009416. doi: 10.1002/14651858.CD009416.pub3. PMID 37306570
- [Result] Donati D, Boccolari P, Giorgi F, Berti L, Platano D, Tedeschi R. Breaking the Cycle of Pain: The Role of Graded Motor Imagery and Mirror Therapy in Complex Regional Pain Syndrome. Biomedicines. 2024 Sep 20;12(9):2140. doi: 10.3390/biomedicines12092140. PMID 39335652
- [Result] Cuenca-Martinez F, Reina-Varona A, Castillo-Garcia J, La Touche R, Angulo-Diaz-Parreno S, Suso-Marti L. Pain relief by movement representation strategies: An umbrella and mapping review with meta-meta-analysis of motor imagery, action observation and mirror therapy. Eur J Pain. 2022 Feb;26(2):284-309. doi: 10.1002/ejp.1870. Epub 2021 Oct 8. PMID 34592050
- [Result] Cacchio A, De Blasis E, De Blasis V, Santilli V, Spacca G. Mirror therapy in complex regional pain syndrome type 1 of the upper limb in stroke patients. Neurorehabil Neural Repair. 2009 Oct;23(8):792-9. doi: 10.1177/1545968309335977. Epub 2009 May 22. PMID 19465507
- [Result] Buraschi, R., Ranica, G., Nicassio, F., Falso, M. V., & Pollet, J. (2024). Efficacy of rehabilitative intervention on pain and function in patients with upper limb complex regional pain syndrome: A systematic review. Topics in Geriatric Rehabilitation, 40(2), 139-146.